

Analysis was conducted using SPSS version 1.0.0.1406. Gender, smoking status, ASA score, and difficulty of surgery were analyzed using Chi-square cross table. Mean duration of total operative time, insufflation time, and mean hospital-stay were analyzed using Student's 2-tailed t-test. The mean intensity of pain was analyzed using Mann-Whitney U test. Inflammatory markers (WBC, Plt, ESR, CRP, Albumin, Cortisol, IL-6, IL-17, TNF- $\alpha$ , IL-1 $\beta$ ) levels were analyzed using Welch's t-test. Subgroup analysis for the inflammatory markers was done to eliminate the effect of dexamethasone given by anesthesia team at the time of anesthesia induction, analysis was done using Welch's t-test. All test set *p*-value was set at 0.05 to consider results significant.